CLINICAL TRIAL: NCT05280262
Title: Biomarkers for Chemotherapy Associated Neurotoxicity
Acronym: BioCAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GN18ON516P
Record Dates: First submitted 2021-09-14; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Chemotherapy-Related Cognitive Impairment
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment

STUDY DESIGN:
Masking Description: No blinding on trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 Asymptomatic (Other): Group 1 - Prospective cohort of children and young adults enrolled at diagnosis and followed longitudinally
  Patients will be evaluated at 5 time-points (Baseline - Follow Up 1-4 [FU1-4]) during therapy using a computer-based short age-appropriate neurocognitive test battery (CogState) and paired CSF samples taken at the time of routine scheduled lumbar punctures. In addition one saliva sample (or stored DNA from a remission bone marrow sample extracted during routine trial procedures) will be collected as a source of germline DNA and a clinical report form will be completed at study entry and at completion of the study. CSF samples will be collected at the time of the patient's scheduled therapeutic treatment with no additional sampling.
  Interventions: Diagnostic Test: CogState Test
- Group 2 Symptomatic (Other): Group 2 - Children and young adults with Stroke-like syndrome/PRES and /or seizures (SPS)
  Following a diagnosis of SPS, patients and their families can be approached for informed consent to enter this study within 4 weeks following SPS event. If consent is obtained, patients will be evaluated at up to 7 timepoints, or until end of treatment, using a computer-based short age-appropriate neurocognitive test battery (CogState) and paired CSF samples taken at the time of routine scheduled lumbar punctures. Follow up visit 2 will take place at 12 months, with Follow up 3-7 [FU3-7] scheduled at 6 monthly timepoints. CSF samples will be collected at the time of the patient's scheduled therapeutic treatment with no additional sampling.
  Interventions: Diagnostic Test: CogState Test

INTERVENTIONS:
Diagnostic Test: CogState Test — Computerized cognitive testing which provides a score/measurement of distinct cognitive functions

SUMMARY:
To assess if biomarkers can be used to predict early treatment related neurotoxicity in patients with Acute lymphoblastic leukaemia (ALL) or lymphoblastic lymphoma (LBL) and to inform development of novel interventions.

DETAILED DESCRIPTION:
Neurotoxicity during treatment for childhood ALL/LBL remains a significant problem. It can be acute as in the "stroke-like syndrome" seen with methotrexate, or may result in chronic neurocognitive defects. Neurocognitive impairment is estimated to occur in between 20-50% of long-term survivors. Although mean effects on global measures such as intelligence quotient (IQ) are moderate, this hides a significant number of severely affected individuals and the risk factors for severe impairment are poorly understood. Recent studies have highlighted that neurocognitive impairment may continue to evolve throughout adulthood, even with chemotherapy-only regimes. Worryingly, reported imaging and neurocognitive results are similar to those seen in early-onset dementia and the burden of neurological late effects may worsen over the next few decades. Thus, there is an urgent need to better understand the pathophysiology of neurotoxicity in childhood ALL/LBL, develop ways of identifying children at risk and to devise new treatments and/or protective measures.

For those without overt neurotoxicity symptoms, identification of patients at risk for poor neurocognitive outcomes might be achieved using early sensitive measures of neurocognition. Long-term follow up studies indicate that children treated for ALL/LBL have particular problems with memory, executive functions, attention and processing speed. Whether these can be picked up early enough to act as a biomarker for long-term adverse outcome is unknown and will be tested in this study. Alternatively, biomarkers in cerebrospinal fluid may indicate high levels of toxic metabolites or biochemical markers of neurological damage that precede neurocognitive effects. The most highly implicated neurotoxic drug is methotrexate. Methotrexate pharmacokinetics do not correlate with neurotoxicity but secondary metabolites such as folate, homocysteine, adenosine and glutamate analogues have been implicated in both acute and chronic toxicity. An animal model of methotrexate neurotoxicity suggests that excitotoxic glutamate analogues may cause neurotoxicity by binding to N-methyl D-aspartate (NMDA) receptors. Importantly, in this pre-clinical model, NMDA antagonists can reverse and/or prevent neurotoxicity when administered concurrently with methotrexate. This raises the possibility that cerebrospinal fluid (CSF) biomarkers will not only identify children at risk of neurotoxicity but also inform therapeutic strategies.

Finally, in the era of personalised medicine an alternative approach is to develop a panel of genetic predictors of neurotoxicity, which can prospectively identify high-risk children prior to any damage. Several candidate polymorphisms for chemotherapy-induced neurotoxicity have been proposed using small cohorts of patients with diverse cancer types. The investigators will test these prospectively in a large standardised patient cohort. In addition, patients exhibiting overt chemotherapy related neurotoxicity such as those with SPS are likely to exhibit the highest hazard ratios for genetic predisposition and therefore their inclusion in this study will strengthen the likelihood of finding clinically relevant and actionable polymorphisms.

Overall, the investigators predict that this study will provide significant insights into potential neurocognitive, biochemical and genetic biomarkers for neurotoxicity and provide strong underpinning science to determine whether NMDA antagonists are suitable for prevention and/or treatment of these potentially devastating neurotoxic effects

ELIGIBILITY:
Group 1 Inclusion Criteria

* Patients aged between 4-25 years inclusive at time of study consent (CogState is not validated for use in children aged <4years).
* New diagnosis of ALL/LBL
* Informed written consent by patient or parent/guardian.

Group 2 Inclusion Criteria - who experience an overt neurotoxic event

* Aged 1-25 at time of neurotoxic event
* Undergoing chemotherapy treatment for ALL/LBL
* Documented central neurological toxicity thought to be related to chemotherapy such as methotrexate stroke-like syndrome (SLS) Posterior reversible encephalopathy syndrome (PRES) or seizures with no clear alternative cause (see exclusion criteria below)
* Informed written consent by patient or parent/guardian

Group 1 Exclusion Criteria

* Documented history of neurodevelopmental disorder prior to the diagnosis of ALL/LBL (e.g. Down syndrome, other chromosomal disorders).
* Significant visual impairment preventing computer use.
* Diagnosis of relapsed or second cancer.
* Active meningitis or seizures less than one month from study enrolment
* Patients whose Baseline line and Follow Up 1-4 [FU1-4] lumbar punctures will not be performed in a study centre

Group 2 Exclusion Criteria

* Patients with cerebral venous sinus thrombosis as a cause of their neurological symptoms
* Patients whose symptoms are due to peripheral neuropathy or myopathy
* Patients with clear cause for neurological event unrelated to chemotherapy neurotoxicity e.g. head injury following trauma, acute meningitis, viral encephalitis with known causative organism, seizures secondary to severe electrolyte imbalance or hypoglycaemia

Ages: 4 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Group 1 - Change in CogState aggregated test score between test points 1 and 4 | 2 years
  measure of cognitive decline over time
Group 1 - Change in CSF Homocysteine levels over time | 2 years
  Downstream metabolite thought to be responsible for neurotoxic effects of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Greater Glasgow and Clyde, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No